CLINICAL TRIAL: NCT06163534
Title: TEMPUS PHOENIX HNSCC STUDY: A Longitudinal Multi-Omic Biomarker Profiling Study of Patients With Head & Neck Squamous Cell Carcinoma (HNSCC)
Brief Title: A Longitudinal Multi-Omic Biomarker Profiling Study of Patients With Head & Neck Squamous Cell Carcinoma (HNSCC)
Status: Recruiting | Type: Observational
Sponsor: Tempus AI (Industry)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: TP-CA-006; Pro00074943 (Other: Advarra)
Record Dates: First submitted 2023-11-07; First posted 2023-12-11 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Head and Neck Squamous Cell Carcinoma
Keywords: Oncology; Biomarkers; Genomic Profiling; HNSCC; Cancer; Observational; Registry; Precision Medicine; NGS
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — Blood and tissue will be collected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Metastatic or unresectable recurrent HNSCC: Up to 500 participants (including primary tumor location of pharynx, larynx, oral cavity and oropharynx) with metastatic or unresectable recurrent HNSCC who are intended for first line immunotherapy or combination therapy. No intervention.

SUMMARY:
The study is a prospective, longitudinal, non-interventional, multicenter study of participants with HNSCC who will have tissue and blood based molecular biomarker profiling during their standard of care treatment.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* Willing and able to provide informed consent
* Histologically- or cytologically-confirmed metastatic or unresectable, recurrent HNSCC unsuitable for local therapies
* Intended for first line anti-PD1 or PDL1 monotherapy or combination therapy
* Must submit tumor tissue sample representative of current disease per laboratory manual

Exclusion Criteria:

* Non-squamous histologies (eg, nasopharynx or salivary gland)
* Relapse or recurrence within 6 months of first line chemotherapy and / or chemoradiotherapy
* Tumors that are PD-L1 negative (CPS <1)
* Clinical evidence of an active second invasive malignancy within <2 years of enrollment with the exception of stable prostate cancer on watchful waiting, in situ cervical cancer, in situ breast carcinoma or localized non-melanoma skin cancers
* Unable to comply with study procedures (i.e., not willing or able to have additional blood samples collected)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This protocol targets patients with metastatic or unresectable, recurrent HNSCC intended for first line immunotherapy or combination therapy.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2028-03-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Explore DNA, RNA, immune and other multiomic biomarkers to better understand prognostic or predictive biomarkers and to inform future research for new relevant biomarkers. | 5 years
  Use NGS, ctNDA assessments, RNA analysis, and other multiomic testing to uncover biomarkers of collected blood and tissue samples that may predict outcomes, identify markers related to disease, identify markers related to mechanism of drug action, and inform future research.

SECONDARY OUTCOMES:
Explore changes in relevant DNA, RNA, immune and multiomic biomarkers in longitudinal blood samples, and diagnostic and progression biopsy samples, to understand real-world outcomes and resistance mechanisms. | 5 years
  Correlate biomarkers of collected blood and tissue samples with standard of care therapy real-world outcomes such as overall survival, progression free survival, time to next treatment, and time to treatment discontinuation.
Explore changes in ctDNA from longitudinal blood samples to assess ctDNA as a response biomarker. | 5 years
  Assess changes in ctNDA of collected blood samples using ctDNA clearance factors such as time to clearance, best overall clearance rate, best confirmed clearance, duration, time to ctDNA recurrence with standard of care therapy real-world outcomes such as overall survival, progression free survival, time to next treatment, and time to treatment discontinuation.

CONTACTS AND LOCATIONS:
Overall Officials: Virginia Rhodes, MD, Study Director — Tempus AI, Inc.
Locations (29):
- United States (28):
  - City of Hope, Duarte, California
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - University of California, Los Angeles, Los Angeles, California
  - Stanford, Palo Alto, California
  - Providence Medical Foundation, Santa Rosa, California
  - Morehouse, Atlanta, Georgia
  - Piedmont Healthcare, Atlanta, Georgia
  - Winship Cancer Institute, Emory University, Atlanta, Georgia
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - Cancer Care Specialists of Illinois, Decatur, Illinois
  - Illinois Cancer Care, Peoria, Illinois
  - University of Kansas, Westwood, Kansas
  - University of Maryland, Baltimore, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Oncology Hematology Associates, Springfield, Missouri
  - Washington University in St. Louis, St Louis, Missouri
  - Mount Sinai Hospital, New York, New York
  - Sanford Fargo, Fargo, North Dakota
  - University of Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Cancer Care Associates of York, York, Pennsylvania
  - Sanford Sioux Falls, Sioux Falls, South Dakota
  - Vanderbilt University, Nashville, Tennessee
  - University of Washington, Seattle, Washington
  - ThedaCare, Appleton, Wisconsin
- Pan American Cancer for Oncology, San Juan, Puerto Rico

REFERENCES:
- [Background] Hsieh RW, Borson S, Tsagianni A, Zandberg DP. Immunotherapy in Recurrent/Metastatic Squamous Cell Carcinoma of the Head and Neck. Front Oncol. 2021 Sep 1;11:705614. doi: 10.3389/fonc.2021.705614. eCollection 2021. PMID 34540672
- [Background] Head and neck cancer - risk factors and prevention. Cancer.Net. Published June 25, 2012. Accessed August 11, 2023. https://www.cancer.net/cancer-types/head-and-neck-cancer/risk-factors-and-prevention
- [Background] Kimple RJ, Harari PM. The prognostic value of HPV in head and neck cancer patients undergoing postoperative chemoradiotherapy. Ann Transl Med. 2015 May;3(Suppl 1):S14. doi: 10.3978/j.issn.2305-5839.2015.01.37. No abstract available. PMID 26046059
- [Background] Ionna F, Bossi P, Guida A, Alberti A, Muto P, Salzano G, Ottaiano A, Maglitto F, Leopardo D, De Felice M, Longo F, Tafuto S, Della Vittoria Scarpati G, Perri F. Recurrent/Metastatic Squamous Cell Carcinoma of the Head and Neck: A Big and Intriguing Challenge Which May Be Resolved by Integrated Treatments Combining Locoregional and Systemic Therapies. Cancers (Basel). 2021 May 14;13(10):2371. doi: 10.3390/cancers13102371. PMID 34069092
- [Background] Samra B, Tam E, Baseri B, Shapira I. Checkpoint inhibitors in head and neck cancer: current knowledge and perspectives. J Investig Med. 2018 Oct;66(7):1023-1030. doi: 10.1136/jim-2018-000743. Epub 2018 Jun 25. PMID 29941547
- [Background] Vermorken JB, Mesia R, Rivera F, Remenar E, Kawecki A, Rottey S, Erfan J, Zabolotnyy D, Kienzer HR, Cupissol D, Peyrade F, Benasso M, Vynnychenko I, De Raucourt D, Bokemeyer C, Schueler A, Amellal N, Hitt R. Platinum-based chemotherapy plus cetuximab in head and neck cancer. N Engl J Med. 2008 Sep 11;359(11):1116-27. doi: 10.1056/NEJMoa0802656. PMID 18784101
- [Background] Burtness B, Harrington KJ, Greil R, Soulieres D, Tahara M, de Castro G Jr, Psyrri A, Baste N, Neupane P, Bratland A, Fuereder T, Hughes BGM, Mesia R, Ngamphaiboon N, Rordorf T, Wan Ishak WZ, Hong RL, Gonzalez Mendoza R, Roy A, Zhang Y, Gumuscu B, Cheng JD, Jin F, Rischin D; KEYNOTE-048 Investigators. Pembrolizumab alone or with chemotherapy versus cetuximab with chemotherapy for recurrent or metastatic squamous cell carcinoma of the head and neck (KEYNOTE-048): a randomised, open-label, phase 3 study. Lancet. 2019 Nov 23;394(10212):1915-1928. doi: 10.1016/S0140-6736(19)32591-7. Epub 2019 Nov 1. PMID 31679945
- [Background] Wang HC, Yeh TJ, Chan LP, Hsu CM, Cho SF. Exploration of Feasible Immune Biomarkers for Immune Checkpoint Inhibitors in Head and Neck Squamous Cell Carcinoma Treatment in Real World Clinical Practice. Int J Mol Sci. 2020 Oct 15;21(20):7621. doi: 10.3390/ijms21207621. PMID 33076306
- [Background] Wei SC, Duffy CR, Allison JP. Fundamental Mechanisms of Immune Checkpoint Blockade Therapy. Cancer Discov. 2018 Sep;8(9):1069-1086. doi: 10.1158/2159-8290.CD-18-0367. Epub 2018 Aug 16. PMID 30115704
- [Background] Darvin P, Toor SM, Sasidharan Nair V, Elkord E. Immune checkpoint inhibitors: recent progress and potential biomarkers. Exp Mol Med. 2018 Dec 13;50(12):1-11. doi: 10.1038/s12276-018-0191-1. PMID 30546008
- [Background] Yu C, Li Q, Zhang Y, Wen ZF, Dong H, Mou Y. Current status and perspective of tumor immunotherapy for head and neck squamous cell carcinoma. Front Cell Dev Biol. 2022 Aug 26;10:941750. doi: 10.3389/fcell.2022.941750. eCollection 2022. PMID 36092724
- [Background] Kong L, Birkeland AC. Liquid Biopsies in Head and Neck Cancer: Current State and Future Challenges. Cancers (Basel). 2021 Apr 14;13(8):1874. doi: 10.3390/cancers13081874. PMID 33919778
- [Background] Mazurek AM, Rutkowski T, Fiszer-Kierzkowska A, Malusecka E, Skladowski K. Assessment of the total cfDNA and HPV16/18 detection in plasma samples of head and neck squamous cell carcinoma patients. Oral Oncol. 2016 Mar;54:36-41. doi: 10.1016/j.oraloncology.2015.12.002. Epub 2016 Jan 11. PMID 26786940
- [Background] Bettegowda C, Sausen M, Leary RJ, Kinde I, Wang Y, Agrawal N, Bartlett BR, Wang H, Luber B, Alani RM, Antonarakis ES, Azad NS, Bardelli A, Brem H, Cameron JL, Lee CC, Fecher LA, Gallia GL, Gibbs P, Le D, Giuntoli RL, Goggins M, Hogarty MD, Holdhoff M, Hong SM, Jiao Y, Juhl HH, Kim JJ, Siravegna G, Laheru DA, Lauricella C, Lim M, Lipson EJ, Marie SK, Netto GJ, Oliner KS, Olivi A, Olsson L, Riggins GJ, Sartore-Bianchi A, Schmidt K, Shih lM, Oba-Shinjo SM, Siena S, Theodorescu D, Tie J, Harkins TT, Veronese S, Wang TL, Weingart JD, Wolfgang CL, Wood LD, Xing D, Hruban RH, Wu J, Allen PJ, Schmidt CM, Choti MA, Velculescu VE, Kinzler KW, Vogelstein B, Papadopoulos N, Diaz LA Jr. Detection of circulating tumor DNA in early- and late-stage human malignancies. Sci Transl Med. 2014 Feb 19;6(224):224ra24. doi: 10.1126/scitranslmed.3007094. PMID 24553385
- [Background] Wang Y, Springer S, Mulvey CL, Silliman N, Schaefer J, Sausen M, James N, Rettig EM, Guo T, Pickering CR, Bishop JA, Chung CH, Califano JA, Eisele DW, Fakhry C, Gourin CG, Ha PK, Kang H, Kiess A, Koch WM, Myers JN, Quon H, Richmon JD, Sidransky D, Tufano RP, Westra WH, Bettegowda C, Diaz LA Jr, Papadopoulos N, Kinzler KW, Vogelstein B, Agrawal N. Detection of somatic mutations and HPV in the saliva and plasma of patients with head and neck squamous cell carcinomas. Sci Transl Med. 2015 Jun 24;7(293):293ra104. doi: 10.1126/scitranslmed.aaa8507. PMID 26109104
- [Background] Ahn SM, Chan JY, Zhang Z, Wang H, Khan Z, Bishop JA, Westra W, Koch WM, Califano JA. Saliva and plasma quantitative polymerase chain reaction-based detection and surveillance of human papillomavirus-related head and neck cancer. JAMA Otolaryngol Head Neck Surg. 2014 Sep;140(9):846-54. doi: 10.1001/jamaoto.2014.1338. PMID 25078109
- [Background] Chan KCA, Woo JKS, King A, Zee BCY, Lam WKJ, Chan SL, Chu SWI, Mak C, Tse IOL, Leung SYM, Chan G, Hui EP, Ma BBY, Chiu RWK, Leung SF, van Hasselt AC, Chan ATC, Lo YMD. Analysis of Plasma Epstein-Barr Virus DNA to Screen for Nasopharyngeal Cancer. N Engl J Med. 2017 Aug 10;377(6):513-522. doi: 10.1056/NEJMoa1701717. PMID 28792880
- [Background] Hamana K, Uzawa K, Ogawara K, Shiiba M, Bukawa H, Yokoe H, Tanzawa H. Monitoring of circulating tumour-associated DNA as a prognostic tool for oral squamous cell carcinoma. Br J Cancer. 2005 Jun 20;92(12):2181-4. doi: 10.1038/sj.bjc.6602635. PMID 15928666
- [Background] Chera BS, Kumar S, Shen C, Amdur R, Dagan R, Green R, Goldman E, Weiss J, Grilley-Olson J, Patel S, Zanation A, Hackman T, Blumberg J, Patel S, Thorp B, Weissler M, Yarbrough W, Sheets N, Mendenhall W, Tan XM, Gupta GP. Plasma Circulating Tumor HPV DNA for the Surveillance of Cancer Recurrence in HPV-Associated Oropharyngeal Cancer. J Clin Oncol. 2020 Apr 1;38(10):1050-1058. doi: 10.1200/JCO.19.02444. Epub 2020 Feb 4. PMID 32017652
- [Background] Aulakh SS, Silverman DA, Young K, Dennis SK, Birkeland AC. The Promise of Circulating Tumor DNA in Head and Neck Cancer. Cancers (Basel). 2022 Jun 16;14(12):2968. doi: 10.3390/cancers14122968. PMID 35740633
- [Background] Liebs S, Eder T, Klauschen F, Schutte M, Yaspo ML, Keilholz U, Tinhofer I, Kidess-Sigal E, Braunholz D. Applicability of liquid biopsies to represent the mutational profile of tumor tissue from different cancer entities. Oncogene. 2021 Aug;40(33):5204-5212. doi: 10.1038/s41388-021-01928-w. Epub 2021 Jul 6. PMID 34230613
- [Background] Russano M, Napolitano A, Ribelli G, Iuliani M, Simonetti S, Citarella F, Pantano F, Dell'Aquila E, Anesi C, Silvestris N, Argentiero A, Solimando AG, Vincenzi B, Tonini G, Santini D. Liquid biopsy and tumor heterogeneity in metastatic solid tumors: the potentiality of blood samples. J Exp Clin Cancer Res. 2020 May 27;39(1):95. doi: 10.1186/s13046-020-01601-2. PMID 32460897
- [Background] Litchfield K, Reading JL, Puttick C, Thakkar K, Abbosh C, Bentham R, Watkins TBK, Rosenthal R, Biswas D, Rowan A, Lim E, Al Bakir M, Turati V, Guerra-Assuncao JA, Conde L, Furness AJS, Saini SK, Hadrup SR, Herrero J, Lee SH, Van Loo P, Enver T, Larkin J, Hellmann MD, Turajlic S, Quezada SA, McGranahan N, Swanton C. Meta-analysis of tumor- and T cell-intrinsic mechanisms of sensitization to checkpoint inhibition. Cell. 2021 Feb 4;184(3):596-614.e14. doi: 10.1016/j.cell.2021.01.002. Epub 2021 Jan 27. PMID 33508232
- [Background] Fairfax BP, Taylor CA, Watson RA, Nassiri I, Danielli S, Fang H, Mahe EA, Cooper R, Woodcock V, Traill Z, Al-Mossawi MH, Knight JC, Klenerman P, Payne M, Middleton MR. Peripheral CD8+ T cell characteristics associated with durable responses to immune checkpoint blockade in patients with metastatic melanoma. Nat Med. 2020 Feb;26(2):193-199. doi: 10.1038/s41591-019-0734-6. Epub 2020 Feb 10. PMID 32042196
- [Background] Valpione S, Galvani E, Tweedy J, Mundra PA, Banyard A, Middlehurst P, Barry J, Mills S, Salih Z, Weightman J, Gupta A, Gremel G, Baenke F, Dhomen N, Lorigan PC, Marais R. Immune-awakening revealed by peripheral T cell dynamics after one cycle of immunotherapy. Nat Cancer. 2020 Feb;1(2):210-221. doi: 10.1038/s43018-019-0022-x. Epub 2020 Feb 10. PMID 32110781
- [Background] Nabet BY, Esfahani MS, Moding EJ, Hamilton EG, Chabon JJ, Rizvi H, Steen CB, Chaudhuri AA, Liu CL, Hui AB, Almanza D, Stehr H, Gojenola L, Bonilla RF, Jin MC, Jeon YJ, Tseng D, Liu C, Merghoub T, Neal JW, Wakelee HA, Padda SK, Ramchandran KJ, Das M, Plodkowski AJ, Yoo C, Chen EL, Ko RB, Newman AM, Hellmann MD, Alizadeh AA, Diehn M. Noninvasive Early Identification of Therapeutic Benefit from Immune Checkpoint Inhibition. Cell. 2020 Oct 15;183(2):363-376.e13. doi: 10.1016/j.cell.2020.09.001. Epub 2020 Oct 1. PMID 33007267
- [Background] Beaubier N, Tell R, Lau D, Parsons JR, Bush S, Perera J, Sorrells S, Baker T, Chang A, Michuda J, Iguartua C, MacNeil S, Shah K, Ellis P, Yeatts K, Mahon B, Taxter T, Bontrager M, Khan A, Huether R, Lefkofsky E, White KP. Clinical validation of the tempus xT next-generation targeted oncology sequencing assay. Oncotarget. 2019 Mar 22;10(24):2384-2396. doi: 10.18632/oncotarget.26797. eCollection 2019 Mar 22. PMID 31040929
- [Background] Beaubier N, Bontrager M, Huether R, Igartua C, Lau D, Tell R, Bobe AM, Bush S, Chang AL, Hoskinson DC, Khan AA, Kudalkar E, Leibowitz BD, Lozachmeur A, Michuda J, Parsons J, Perera JF, Salahudeen A, Shah KP, Taxter T, Zhu W, White KP. Integrated genomic profiling expands clinical options for patients with cancer. Nat Biotechnol. 2019 Nov;37(11):1351-1360. doi: 10.1038/s41587-019-0259-z. Epub 2019 Sep 30. PMID 31570899
- [Background] Finkle JD, Boulos H, Driessen TM, Lo C, Blidner RA, Hafez A, Khan AA, Lozac'hmeur A, McKinnon KE, Perera J, Zhu W, Dowlati A, White KP, Tell R, Beaubier N. Validation of a liquid biopsy assay with molecular and clinical profiling of circulating tumor DNA. NPJ Precis Oncol. 2021 Jul 2;5(1):63. doi: 10.1038/s41698-021-00202-2. PMID 34215841